CLINICAL TRIAL: NCT04234191
Title: Comparing Rapid Micro-Induction and Standard Induction of Buprenorphine/Naloxone for Treatment of Opioid Use Disorder: A Randomized Controlled Trial
Brief Title: Comparing Rapid Micro-Induction and Standard Induction of Buprenorphine/Naloxone for Treatment of Opioid Use Disorder
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Vancouver Coastal Health (Other Government)
Responsible Party: Principal Investigator, Nickie Mathew, Clinical Associate Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H19-03254
Record Dates: First submitted 2020-01-13; First posted 2020-01-21 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Opioid Use Disorder
Keywords: Buprenorphine/naloxone; Suboxone; Opioid agonist treatment; Micro-induction; Microdosing; Withdrawal Management
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine, Naloxone Drug Combination; Hydromorphone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Rapid Micro-Induction (Experimental): On Day 1, participants will receive 0.5mg bup/nx sublingually (SL) every 3 hours (Q3H) - total daily dose of 4mg. On Day 2, they will receive 1mg bup/nx SL Q3H - total daily dose of 8mg. On Day 3, they will receive 8mg bup/nx SL once and 1-4mg bup/nx SL Q3H as needed (PRN) for withdrawal symptoms and/or craving and/or pain - maximum daily dose of 32mg. Afterwards, their day 3 total dose will be consolidated to once daily dosing - maximum daily dose of 32mg. On Days 1 and 2, participants will concurrently receive 1-48mg hydromorphone orally, intravenously, subcutaneously, or intramuscularly (PO/IV/SC/IM) Q1 to 3H PRN for withdrawal symptoms and/or craving and/or pain, titrated to effect (start at lower end of dosing range). Hydromorphone will be discontinued on Days 3 onwards.
  Interventions: Drug: Buprenorphine/naloxone; Drug: Hydromorphone
- Standard Induction (Active Comparator): Day 1 is initiated when participants score 11 or above on the Clinical Opiate Withdrawal Scale (COWS), and when they have been abstinent from short-acting opioids for at least 6-12 hours or from long-acting opioids for 24-72 hours. On Day 1, participants will start with 2 or 4mg bup/nx SL. If their COWS score increases, bup/nx will be held. If their COWS score remains the same or decreases, additional dosing can be done in increments of 2mg bup/nx SL every 2 hours (Q2H) as needed (PRN). On Day 2, dosing will be consolidated to once daily dosing. The maximum total daily dose for Day 1 and 2 is 32mg.
  Interventions: Drug: Buprenorphine/naloxone

INTERVENTIONS:
Drug: Buprenorphine/naloxone — Buprenorphine/naloxone is an opioid agonist treatment for opioid use disorder. It is administered via sublingual tablet form.
  Other Names: Suboxone
Drug: Hydromorphone — Hydromorphone is an opioid used for managing pain, craving, and withdrawal. It is administered orally via tablet or liquid form; or administered intravenously, subcutaneously, or intramuscularly via liquid form.
  Other Names: Dihydromorphinone, Dilaudid
  Arms: Rapid Micro-Induction

SUMMARY:
The current first-line treatment for opioid use disorder (OUD) in Canada is buprenorphine/naloxone (bup/nx). The standard induction method of bup/nx requires patients to be abstinent from opioids and thereby experience withdrawal symptoms prior to induction, which can be a major barrier in starting treatment. Rapid micro-induction (also known as micro-dosing, low-dose induction) involves the administration of small, frequent does of bup/nx and removes the need for a period of withdrawal prior to the start of treatment. This study aims to compare the effectiveness and safety of rapid micro-induction versus standard induction of bup/nx in patients with OUD.

DETAILED DESCRIPTION:
This is a randomized, controlled, open-label superiority trial involving 50 individuals with OUD. Participants will be randomized into two arms: rapid micro-induction and standard induction (based on the American Society of Addiction Medicine Practice Guidelines and product monograph) of bup/nx.

ELIGIBILITY:
Inclusion Criteria:

1. Opioid Use Disorder (OUD) as defined by the Diagnostic and Statistical Manual of Mental Disorders-5 diagnostic criteria;
2. Individuals seeking Opioid Agonist Treatment (OAT);
3. Be 19 years of age or older;
4. Be willing and able to adhere to the study protocol and follow-up schedule;
5. Be able to provide written informed consent to participate in the clinical trial.
6. If female and of childbearing potential, agree to use an effective method of birth control approved by the study investigators throughout the study.

Exclusion Criteria:

1. Diagnosis of severe medical or psychiatric conditions contraindicated for buprenorphine/naloxone or hydromorphone treatment;
2. Anticipated deterioration of health due to discontinuation of medications that are contraindicated with buprenorphine/naloxone and/or hydromorphone;
3. Positive pregnancy test for women of childbearing potential;
4. Methadone use in the past 5 days;
5. Buprenorphine use in the past 5 days;
6. Known allergy or sensitivity to buprenorphine/naloxone and/or hydromorphone;
7. Anticipation that the patient may need to initiate pharmacological treatment during the trial that is deemed unsafe by the study physician or could prevent study completion;
8. Unwilling or unable to use an effective method of birth control approved by the study investigators throughout the study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-08-18 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Successful induction of bup/nx with low levels of withdrawal | Baseline to Day 1 (Standard Induction Arm) or Day 2 (Rapid Micro-Induction Arm)
  This is defined as the following: participants who remain in treatment until they have received a total daily dose of ≥ 8mg of bup/nx (successful induction), and score ≤ 12 on the COWS (low levels of withdrawal) from baseline to when they reach that dose.

SECONDARY OUTCOMES:
Illicit drug use | Baseline to Day 1 (Standard Induction Arm) or Day 2 (Rapid Micro-Induction Arm)
  Assessed by urine drug screens (UDS) and Treatment Outcomes Profile (TOP).
Drug use behaviour | Baseline to Day 1 (Standard Induction Arm) or Day 2 (Rapid Micro-Induction Arm)
  Assessed by the Treatment Outcomes Profile (TOP).
Treatment retention | Day 7
  Participants who pick up their prescription of bup/nx on Day 7. Assessed via the pharmacy database.
Craving | Baseline to Day 1 (Standard induction Arm) or Day 2 (Rapid Micro-Induction Arm)
  Assessed by the numeric craving scale.
Pain | Baseline to Day 1 (Standard induction Arm) or Day 2 (Rapid Micro-Induction Arm)
  Assessed by the numeric pain scale.
Physical health | Baseline (both arms)
  Assessed by the health section of the Opiate Treatment Index (OTI).
Client satisfaction | Day 1 (Standard induction Arm) or Day 2 (Rapid Micro-Induction Arm)
  Assessed by the Treatment Perceptions Questionnaire (TPQ).
Appearance of adverse events | Baseline to Day 1 (Standard induction Arm) or Day 2 (Rapid Micro-Induction Arm)
  Assessed by an adverse events report form.

CONTACTS AND LOCATIONS:
Overall Officials: Pouya Azar, MD, FRCPC, DABAM, Principal Investigator — University of British Columbia; Nickie Mathew, MD, MSc, FRCPC, ABPN, ABPM, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.

REFERENCES:
- [Background] Sandhu R, Zivanovic R, Klaire S, Nikoo M, Rozylo J, Azar P. Buprenorphine/naloxone induction for treatment of acute on chronic pain using a micro-dosing regimen: A case report. Can J Pain. 2019 Apr 25;3(1):79-84. doi: 10.1080/24740527.2019.1599279. eCollection 2019. PMID 35005396
- [Background] Klaire S, Zivanovic R, Barbic SP, Sandhu R, Mathew N, Azar P. Rapid micro-induction of buprenorphine/naloxone for opioid use disorder in an inpatient setting: A case series. Am J Addict. 2019 Jul;28(4):262-265. doi: 10.1111/ajad.12869. Epub 2019 Mar 22. PMID 30901127
- [Background] Hammig R, Kemter A, Strasser J, von Bardeleben U, Gugger B, Walter M, Dursteler KM, Vogel M. Use of microdoses for induction of buprenorphine treatment with overlapping full opioid agonist use: the Bernese method. Subst Abuse Rehabil. 2016 Jul 20;7:99-105. doi: 10.2147/SAR.S109919. eCollection 2016. PMID 27499655
- [Background] Vogel M, Kock P, Strasser J, Wiesbeck G, Walter M, Dursteler KM. Chronic High-Dose Buprenorphine Does Not Block Subjective High from Diacetylmorphine in a Patient in Heroin-Assisted Treatment. J Psychoactive Drugs. 2019 Sep-Oct;51(4):377-382. doi: 10.1080/02791072.2019.1610200. Epub 2019 May 2. PMID 31046631
- [Background] Kampman K, Jarvis M. American Society of Addiction Medicine (ASAM) National Practice Guideline for the Use of Medications in the Treatment of Addiction Involving Opioid Use. J Addict Med. 2015 Sep-Oct;9(5):358-67. doi: 10.1097/ADM.0000000000000166. PMID 26406300
- [Derived] Wong JSH, Nikoo M, Westenberg JN, Suen JG, Wong JYC, Krausz RM, Schutz CG, Vogel M, Sidhu JA, Moe J, Arishenkoff S, Griesdale D, Mathew N, Azar P. Comparing rapid micro-induction and standard induction of buprenorphine/naloxone for treatment of opioid use disorder: protocol for an open-label, parallel-group, superiority, randomized controlled trial. Addict Sci Clin Pract. 2021 Feb 12;16(1):11. doi: 10.1186/s13722-021-00220-2. PMID 33579359